CLINICAL TRIAL: NCT02659319
Title: Intervening in Family and Peer Contexts to Decrease Child Overweight
Brief Title: Families and Schools for Health
Acronym: FiSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amanda Harrist (Other)
Responsible Party: Sponsor-Investigator, Amanda Harrist, Professor, Oklahoma State University
Organization: Oklahoma State University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: NIFA/USDA Agreement No. 05545; HR07-044, HR08-043 (Other Grant/Funding Number: Oklahoma Health Research Program)
Record Dates: First submitted 2016-01-07; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Overweight; Pediatric Obesity
Keywords: Child overweight; Child obesity; Family dynamics; Peer relationships; Family intervention; School intervention; Parenting
MeSH Terms: conditions — Overweight; Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Family Lifestyle (FL; n = 117) (Experimental): This arm includes the Family Food & Lifestyle intervention (FL). Parents and children meet for 12 weekly, 90-minute psychoeducational groups in children's schools. They meet separately for 45 minutes and then conjointly for 45 minutes.
  Interventions: Behavioral: Family Lifestyle (FL)
- FL + Family Dynamics (FL+FD; n = 88) (Experimental): This arm includes the Family Food & Lifestyle + Family Dynamics interventions (FL+FD). Parents and children meet separately for the full 90-minute psychoeducation sessions. The first 45 minutes are devoted to the Family Food & Lifestyle intervention and the second 45 minutes to the Family Dynamics intervention.
  Interventions: Behavioral: Family Lifestyle (FL); Behavioral: Family Dynamics (FD)
- FL + Peer Group (FL+PG; n = 124) (Experimental): This arm includes the Family Food & Lifestyle intervention plus the 12-session, Peer Group intervention.
  Interventions: Behavioral: Family Lifestyle (FL); Behavioral: Peer Group (PG)
- FL + FD + Peer Group (FL+FD+PG; n = 130) (Experimental): This arm includes the Family Food & Lifestyle intervention plus the Family Dynamics Intervention plus the Peer Group intervention.
  Interventions: Behavioral: Family Lifestyle (FL); Behavioral: Family Dynamics (FD); Behavioral: Peer Group (PG)
- Control (n = 82) (No Intervention): Non-intervention control group

INTERVENTIONS:
Behavioral: Family Lifestyle (FL) — 12-week Family Food & Lifestyle intervention, aimed at improving family nutritional intake, activity levels, weight perception, and parental monitoring of child eating. Material is delivered in psychoeducational groups in the children's schools.
  Arms: FL + FD + Peer Group (FL+FD+PG; n = 130); FL + Family Dynamics (FL+FD; n = 88); FL + Peer Group (FL+PG; n = 124); Family Lifestyle (FL; n = 117)
Behavioral: Family Dynamics (FD) — The Family Dynamics intervention focuses on positive parenting (i.e., emotion coaching, praise, limit setting) and on child emotion regulation and positive problem solving. Material is delivered in psychoeducational groups in the children's schools.
  Arms: FL + FD + Peer Group (FL+FD+PG; n = 130); FL + Family Dynamics (FL+FD; n = 88)
Behavioral: Peer Group (PG) — Peer Group intervention conducted throughout one semester of the school year that includes 12 sessions of a guidance-type curriculum during class time sensitizing children to the importance of social inclusion of all children
  Arms: FL + FD + Peer Group (FL+FD+PG; n = 130); FL + Peer Group (FL+PG; n = 124)

SUMMARY:
The purpose of the study is to test the effectiveness of a child obesity intervention with multiple components targeting nutrition and/or psycho-social factors in children, their parents, and their classmates. The specific aims of the study are to (1) Determine the effectiveness of two family-level interventions for improving child outcomes (unhealthy eating, low activity, and overweight); (2) Determine the extent to which adding a family dynamics component enhances the effectiveness of a family lifestyle intervention and improves the child outcomes listed above; and (3) Determine the extent to which a peer-level intervention improves the effectiveness of two family-level interventions among overweight children.

DETAILED DESCRIPTION:
The Families and Schools for Health (FiSH) Project evaluates a psychosocial intervention that targets the family and peer contexts of overweight children. 23 rural schools were identified for participation (schools within a 90-mile radius of the PI's campus were targeted) and each was assigned to one of five intervention conditions using stratified random sampling, with stratification based on proximity to each other (to avoid spill-over effects) and proportion of Native American Indian students. A community sample of 1186 1st grade children, their families, and their teachers were successfully recruited. Anthropometric assessments were conducted with the 1186 children. Those who were not at Control schools were invited to participate in the intervention. 541 children qualified for the intervention (i.e., had BMI% > 75%), including 459 at Intervention schools and 82 at Control schools. Intervention conditions were (1) a 12-week Family Food & Lifestyle intervention (FL), aimed at improving family nutritional intake, activity levels, weight perception, and parental monitoring of child eating; (2) a 12-week Family Food & Lifestyle and Family Dynamics intervention (FL+FD) that additionally targets dysfunctional family patterns such as high conflict, poor parent-child communication, and parental over-control or permissiveness; and (3) a Peer Group (PG) intervention conducted throughout one semester of the school year that includes a guidance-type curriculum sensitizing children to the importance of social inclusion of all children. Thus, 5 treatment groups were evaluated in the intervention year and followed through 4th grade: FL, FL+FD, FL+PG, FL+FD+PG, and Control. Child psychosocial variables such as emotional eating, self-esteem, loneliness, and social withdrawal will be analyzed as mediators between family/peer contexts and child overweight.

ELIGIBILITY:
Inclusion Criteria:

* Children with BMI% greater than or equal to 75% who were enrolled in first grade in participating schools.

Exclusion Criteria:

* Children with BMI% < 75%.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2005-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Body Mass Change from Baseline to End of 1st grade | Wave 2, Spring Year 1
  Height and weight measured at Wave 2 (Spring 1st grade), vs. Baseline at Fall 1st grade
Body Mass Change from Baseline to End of 2nd grade | Wave 3, Spring Year 2
  Height and weight measured at Wave 3 (Spring 2nd grade), vs. Baseline at Wave 1, Fall 1st grade
Body Mass Change from Baseline to End of 3rd grade | Wave 4, Spring Year 3
  Height and weight measured at Wave 4 (Spring 3rd grade), vs. Baseline at Wave 1, Fall 1st grade
Body Mass Change from Baseline to End of 4th grade | Wave 5, Spring Year 4
  Height and weight measured at Wave 5 (Spring 4th grade) vs. Baseline at Wave 1, Fall 1st grade

SECONDARY OUTCOMES:
Parent perceived responsibility, weight, child weight, concerns about weight, feeding practices - parent report | Wave 1 Fall year 1, Wave 2 Spring year 1, Wave 3 Spring year 2, Wave 4 Spring year 3, Wave 5 Spring year 4
Parent expectations about, parent modeling of, and parent perception of child beliefs regarding eating - parent report | Wave 1 Fall year 1, Wave 2 Spring year 1, Wave 3 Spring year 2, Wave 4 Spring year 3, Wave 5 Spring year 4
Family problem solving, communication, affective responsiveness, affective involvement, & general family functioning - parent report | Wave 1 Fall year 1, Wave 2 Spring year 1, Wave 3 Spring year 2, Wave 4 Spring year 3, Wave 5 Spring year 4
Parenting style (permissive, authoritative, authoritarian) - parent report | Wave 1 Fall year 1, Wave 2 Spring year 1, Wave 3 Spring year 2, Wave 4 Spring year 3, Wave 5 Spring year 4
Parent response to child negative emotions - parent report | Wave 1 Fall year 1, Wave 2 Spring year 1, Wave 3 Spring year 2, Wave 4 Spring year 3, Wave 5 Spring year 4
Child temperament - child and parent report | Wave 2 Spring year 1, Wave 3 Spring year 2, Wave 4 Spring year 3, Wave 5 Spring year 4
Child emotion management - Parent and child report | Wave 2 Spring year 1, Wave 3 Spring year 2, Wave 4 Spring year 3, Wave 5 Spring year 4
Child behavior problems - Parent and teacher report (externalizing, internalizing) | Wave 1 Fall year 1, Wave 2 Spring year 1, Wave 3 Spring year 2, Wave 4 Spring year 3, Wave 5 Spring year 4
School climate | Wave 1 Fall year 1, Wave 2 Spring year 1, Wave 3 Spring year 2, Wave 4 Spring year 3, Wave 5 Spring year 4
Peer relations - child, peer, and teacher reports | Wave 1 Fall year 1, Wave 2 Spring year 1, Wave 3 Spring year 2, Wave 4 Spring year 3, Wave 5 Spring year 4
Child emotional and external eating - child self report | Wave 1 Fall year 1, Wave 2 Spring year 1, Wave 3 Spring year 2, Wave 4 Spring year 3, Wave 5 Spring year 4
Body esteem - child self report | Wave 1 Fall year 1, Wave 2 Spring year 1, Wave 3 Spring year 2, Wave 4 Spring year 3, Wave 5 Spring year 4
Child self esteem - child self report | Wave 1 Fall year 1, Wave 2 Spring year 1, Wave 3 Spring year 2, Wave 4 Spring year 3, Wave 5 Spring year 4
Child depressive symptoms - child self report | Wave 1 Fall year 1, Wave 2 Spring year 1, Wave 3 Spring year 2, Wave 4 Spring year 3, Wave 5 Spring year 4

CONTACTS AND LOCATIONS:
Overall Officials: Amanda W Harrist, PhD, Principal Investigator — Oklahoma State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harrist AW, Swindle TM, Hubbs-Tait L, Topham GL, Shriver LH, Page MC. The Social and Emotional Lives of Overweight, Obese, and Severely Obese Children. Child Dev. 2016 Sep;87(5):1564-80. doi: 10.1111/cdev.12548. Epub 2016 May 25. PMID 27223340
- [Background] Shriver LH, Hubbs-Tait L, Harrist AW, Topham G, Page M. Child gender and weight status moderate the relation of maternal feeding practices to body esteem in 1st grade children. Appetite. 2015 Jun;89:62-9. doi: 10.1016/j.appet.2015.01.017. Epub 2015 Jan 23. PMID 25624022
- [Background] Harrist AW, Hubbs-Tait L, Topham GL, Shriver LH, Page MC. Emotion regulation is related to children's emotional and external eating. J Dev Behav Pediatr. 2013 Oct;34(8):557-65. doi: 10.1097/DBP.0b013e3182a5095f. PMID 24131878
- [Background] Shriver LH, Harrist AW, Page M, Hubbs-Tait L, Moulton M, Topham G. Differences in body esteem by weight status, gender, and physical activity among young elementary school-aged children. Body Image. 2013 Jan;10(1):78-84. doi: 10.1016/j.bodyim.2012.10.005. Epub 2012 Nov 24. PMID 23228485
- [Background] Harrist, A. W., Topham, G. L., Hubbs-Tait, L., Page, M. C., Kennedy, T. S., & Shriver, L. H. (2012). What developmental science can contribute to a multidisciplinary understanding of childhood obesity. Child Development Perspectives, 6, 445-465. doi:10.1111/cdep.12004
- [Background] Shriver LH, Harrist AW, Hubbs-Tait L, Topham G, Page M, Barrett A. Weight status, physical activity, and fitness among third-grade rural children. J Sch Health. 2011 Sep;81(9):536-44. doi: 10.1111/j.1746-1561.2011.00624.x. PMID 21831066
- [Background] Topham GL, Hubbs-Tait L, Rutledge JM, Page MC, Kennedy TS, Shriver LH, Harrist AW. Parenting styles, parental response to child emotion, and family emotional responsiveness are related to child emotional eating. Appetite. 2011 Apr;56(2):261-4. doi: 10.1016/j.appet.2011.01.007. Epub 2011 Jan 11. PMID 21232566
- [Background] Topham GL, Page MC, Hubbs-Tait L, Rutledge JM, Kennedy TS, Shriver L, Harrist AW. Maternal depression and socio-economic status moderate the parenting style/child obesity association. Public Health Nutr. 2010 Aug;13(8):1237-44. doi: 10.1017/S1368980009992163. Epub 2009 Dec 8. PMID 19968899
- [Background] Hubbs-Tait L, Kennedy TS, Page MC, Topham GL, Harrist AW. Parental feeding practices predict authoritative, authoritarian, and permissive parenting styles. J Am Diet Assoc. 2008 Jul;108(7):1154-61; discussion 1161-2. doi: 10.1016/j.jada.2008.04.008. PMID 18589022